CLINICAL TRIAL: NCT03837119
Title: Maternal and Perinatal Pregnancy Outcome in Women With Heterozygous Hemoglobinopathies
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00101; sp19Hoesli
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2021-06

CONDITIONS: Heterozygous Haemoglobinopathy
Keywords: pregnancy; gestational diabetes; cholestasis in pregnancy; urinary tract infection in pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Pregnancy Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heterozygous Hemoglobinopathy: pregnancy outcome in women with heterozygous hemoglobinopathy
  Interventions: Other: pregnancy outcome
- No Heterozygous Hemoglobinopathy: pregnancy outcome in women without heterozygous hemoglobinopathy
  Interventions: Other: pregnancy outcome

INTERVENTIONS:
Other: pregnancy outcome — descriptive statistics of variables

SUMMARY:
This retrospective study aims to investigate pregnancy outcome in women with heterozygous hemoglobinopathies (regarding gestational diabetes, cholestasis and urinary tract infections) and to analyze if there are aggravated maternal and/or perinatal risks.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with or without heterozygous hemoglobinopathy

Exclusion Criteria:

* refusal of study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women being treated at Universitätsspital Basel/ Frauenklinik (from 2015 until 2017) and at Universitätsspital Zürich (from 2004-2006)
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
gestational diabetes | in the course of pregnancy until delivery
  number of women developing gestational diabetes in pregnancy
cholestasis in pregnancy | in the course of pregnancy until delivery
  number of women developing cholestasis in pregnancy
urinary tract infection | in the course of pregnancy until delivery
  number of women developing urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hoesli, Prof. Dr. MD, Principal Investigator — Frauenklinik Universitätsspital Basel
Locations (2):
- Switzerland (2):
  - Frauenklinik University Hospital Basel, Basel
  - Frauenklinik University Hospital Zürich, Zurich

REFERENCES:
- [Result] Kasparek J, Burkhardt T, Hoesli I, Amstad Bencaiova G. Pregnancy outcomes in women with a hemoglobinopathy trait: a multicenter, retrospective study. Arch Gynecol Obstet. 2021 Nov;304(5):1197-1203. doi: 10.1007/s00404-021-06058-y. Epub 2021 Apr 11. PMID 33842991